CLINICAL TRIAL: NCT02971228
Title: The Bionic Pancreas Feasibility Trial Testing the Bionic Pancreas With ZP4207
Brief Title: Feasibility Trial Testing the Bionic Pancreas With ZP4207
Acronym: dasiglucagon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Massachusetts General Hospital (Other); Beta Bionics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZP4207-16051
Record Dates: First submitted 2016-11-03; First posted 2016-11-22 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: glucagon; Type 1 diabetes mellitus; Bionic Pancreas; diabetes; iLet; iPhone; Beta Bionics; Anti-hypoglycemia; Glucagon Analog
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin Lispro; dasiglucagon; Glucagon; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1, Lilly glucagon then ZP4207 (Experimental): In Part 1, 12 patients participated in 1-day treatment arms in random order (iPhone-based Bionic Pancreas using Lilly glucagon and iPhone-based Bionic Pancreas using ZP4207 (dasiglucagon) {experimental drug} with insulin lispro) according to pre-generated randomization scheme.
  Interventions: Drug: Insulin Lispro; Drug: ZP4207 (dasiglucagon); Drug: Glucagon; Device: iPhone-based bionic pancreas
- Part 1, ZP4207 then Lilly Glucagon (Experimental): In Part 1, 12 patients participated in 1-day treatment arms in random order (iPhone-based Bionic Pancreas using Lilly glucagon and iPhone-based Bionic Pancreas using ZP4207 (dasiglucagon) {experimental drug} with insulin lispro) according to pre-generated randomization scheme.
  Interventions: Drug: Insulin Lispro; Drug: ZP4207 (dasiglucagon); Drug: Glucagon; Device: iPhone-based bionic pancreas
- Part 2, Lilly glucagon then ZP4207 (Experimental): In Part 2, it was planned to enrol up to 10 new patients to participate in 1-day treatment arms in random order (iLet-based Bionic Pancreas using Lilly glucagon and iLet-based Bionic Pancreas using ZP4207 (dasiglucagon) {experimental drug} with insulin lispro) according to pre-generated randomization scheme. However, due to unavailability of the iLet, the sponsor decided to stop the trial upon completion of Part 1. Part 2 of the trial using the iLet was consequently not conducted.
  Interventions: Drug: Insulin Lispro; Drug: ZP4207 (dasiglucagon); Drug: Glucagon; Device: iLet-based bionic pancreas
- Part 2, ZP4207 then Lilly Glucagon (Experimental): In Part 2, it was planned to enrol up to 10 new patients to participate in 1-day treatment arms in random order (iLet-based Bionic Pancreas using Lilly glucagon and iLet-based Bionic Pancreas using ZP4207 (dasiglucagon) {experimental drug} with insulin lispro) according to pre-generated randomization scheme. However, due to unavailability of the iLet, the sponsor decided to stop the trial upon completion of Part 1. Part 2 of the trial using the iLet was consequently not conducted.
  Interventions: Drug: Insulin Lispro; Drug: ZP4207 (dasiglucagon); Drug: Glucagon; Device: iLet-based bionic pancreas

INTERVENTIONS:
Drug: Insulin Lispro — Used to lower blood glucose. Commercially available by prescription and is indicated for patients with type 1 diabetes mellitus (T1DM), but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  Other Names: HumaLOG; HumaLOG Cartridge; HumaLOG KwikPen
Drug: ZP4207 (dasiglucagon) — A glucagon analog not yet approved by the FDA. Subcutaneous administration in one BP arm.
  Other Names: dasiglucagon
Drug: Glucagon — A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  Other Names: Glucagon for injection (rDNA original)
Device: iPhone-based bionic pancreas — An experimental device.
  Arms: Part 1, Lilly glucagon then ZP4207; Part 1, ZP4207 then Lilly Glucagon
Device: iLet-based bionic pancreas — An experimental device.
  Arms: Part 2, Lilly glucagon then ZP4207; Part 2, ZP4207 then Lilly Glucagon

SUMMARY:
The purpose of this study was to determine whether the Bionic Pancreas with ZP4207 (dasiglucagon*) was feasible to improve glycemic control in adults with type 1 diabetes mellitus.

*dasiglucagon is the proposed International Nonproprietary Name (pINN) for ZP4207

DETAILED DESCRIPTION:
This was a single-center, open-label, 2-part, randomized cross-over trial. The trial was to enrol up to 20 adult patients with type 1 diabetes mellitus and assess the safety and efficacy of the Bionic Pancreas (BP) using either the iLet or iPhone platform when used with the glucagon analogue ZP4207 (dasiglucagon) versus Lilly glucagon.

In Part 1, patients participated in two 1-day treatment arms in random order (iPhone-based BP using ZP4207 (dasiglucagon) and iPhone-based BP using Lilly glucagon) according to a pre-generated randomization scheme. In Part 2, it was planned to enrol additional patients to participate in two 1-day treatment arms in random order (iLet using ZP4207 (dasiglucagon) and iLet using Lilly glucagon) according to a pre-generated randomization scheme. However, due to unavailability of the iLet, the sponsor decided to stop the trial upon completion of Part 1. Part 2 of the trial using the iLet was consequently not conducted.

One day the BP will use glucagon analogue ZP4207 (dasiglucagon) and the other day the BP will use Lilly glucagon. Subjects will also receive insulin lispro through the BP on both days. The trial will be conducted at single center, the Massachusetts General Hospital Diabetes Center in Boston, MA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T1DM for at least 1 year, as defined by the American Diabetes Association
2. Age ≥ 18 years
3. Prescription medication regimen stable for >1 month (except for medications not expected to affect trial safety or outcome, in the judgment of the investigator)
4. Diabetes managed using an insulin pump for >=6 months
5. Patients in good health according to age (medical history, physical examination, vital signs, 12-lead electrocardiograms [ECGs], laboratory assessments), as judged by the Investigator

Exclusion Criteria:

1. Previous exposure to ZP4207 or adverse reaction to glucagon
2. History of liver disease or current abnormal liver function tests (LFTs)
3. Renal failure
4. Anemia
5. History of coronary artery disease or congestive heart failure (class III or IV)
6. History of transient ischemic attack or stroke
7. Seizure disorder
8. Cystic fibrosis, pancreatitis, or any other pancreatic disease besides T1DM
9. Other endocrine disorders
10. Use of oral anti-diabetic medications
11. Electronically powered implants
12. Hypertension (≥160/100 mm Hg despite treatment)
13. Inadequate venous (vein) access as determined by trial nurse or physician at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05-24 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1, it was planned to enrol 10 patients in two 1-day treatment arms in random order (iPhone-based bionic pancreas using ZP4207 or Lilly Glucagon) according to a pre-generated randomization scheme. The trial had a crossover design. In all, 19 patients were screened and 13 were randomized, but 1 patient withdrew before treatment. Thus, 12 patients were randomized and treated.
Pre-assignment Details: Part 2 was designed to enroll up to 10 new patients in two 1-day treatment arms in random order (iLet using ZP4207 or Lilly Glucagon). However, due to unavailability of the iLet, the sponsor decided to stop the trial upon completion of Part 1. Part 2 of the trial using the iLet was consequently not conducted.
Groups:
- Part 1 Lilly Glucagon or ZP4207: 1 patient was enrolled but withdrew prior to treatment with either trial drug
- Part 1, Lilly Glucagon Then ZP4207: 7 patients received Lilly Glucagon then ZP4207 in this treatment sequence (2 withdrew before receiving ZP4207). Insulin Lispro was also administered in both treatment arms.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration.
  iPhone-based bionic pancreas: An experimental device.
- Part 1, ZP4207 Then Lilly Glucagon: 5 patients received ZP4207 then Lilly Glucagon in this treatment sequence. Insulin Lispro was also administered in both treatment arms.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration.
  iPhone-based bionic pancreas: An experimental device.
- Part 2, ZP4207 Then Lilly Glucagon; Part 2, Lilly Glucagon Then ZP4207: Part 2 of the trial was not conducted - see above.
Period: Overall Study
Arm/Group | Part 1 Lilly Glucagon or ZP4207 | Part 1, Lilly Glucagon Then ZP4207 | Part 1, ZP4207 Then Lilly Glucagon | Part 2, ZP4207 Then Lilly Glucagon | Part 2, Lilly Glucagon Then ZP4207
Started (Enrolled) | 1 | 7 | 5 | 0 (Due to iLet unavailability, trial was stopped upon completion of Part 1. Part 2 was not conducted.) | 0 (Due to iLet unavailability, trial was stopped upon completion of Part 1. Part 2 was not conducted.)
Randomized and Treated | 0 | 7 | 5 | 0 | 0
Completed | 0 | 5 | 5 | 0 (Due to iLet unavailability, trial was stopped upon completion of Part 1. Part 2 was not conducted.) | 0 (Due to iLet unavailability, trial was stopped upon completion of Part 1. Part 2 was not conducted.)
Not Completed | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Logistical challenges | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the crossover nature of the trial, demographic and baseline characteristics are summarized for the overall population.
Groups:
- Part 1, All Participants: In Part 1, 12 patients participated in 1-day treatment arms in random order (iPhone-based Bionic Pancreas using Lilly glucagon and iPhone-based Bionic Pancreas using ZP4207 (dasiglucagon) {experimental drug} with insulin lispro) according to pre-generated randomization scheme. Note: 13 patients were enrolled and 1 patient withdrew prior to treatment with either trial drug; thus, 12 patients were randomized and treated.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration in one BP arm.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (18.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Body weight [Mean (Standard Deviation); unit: kg] | 80.28 (18.357)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.36 (5.301)
Diabetes duration [Mean (Standard Deviation); unit: years] | 28.2 (14.72)
HbA1c [Mean (Standard Deviation); unit: %] | 7.18 (1.462)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Measured by Adverse Events, Local Tolerability of Infusion Site Reactions, and Clinical Laboratory Parameters
Description: Safety and tolerability of ZP4207 in the BP using either the iPhone or the iLet platform, as measured by adverse events (AEs), local tolerability of infusion site reactions, and clinical laboratory parameters.
  See adverse events section for results on AEs by system organ class and preferred term. Clinical laboratory parameters in terms of overall 'investigations' AEs and abnormal hematology parameters that did not resolve by the follow-up visit are presented below. LLN = lower limit of the normal range. Investigations and vital signs AEs by preferred term are presented in the AE section.
  Participants with infusion site pain and nausea measured by visual analog scales (VAS) are presented below; mean values are presented under secondary outcomes. For the VAS, individuals marked on a 10-cm line corresponding to the amount of pain or nausea being experienced, with low scores (cm) indicating no feelings of pain or nausea and high scores (cm) indicating high feelings of pain or nausea.
Time Frame: Up to 50 days
Population: The full analysis set (intent-to-treat population) consisted of all randomized patients: 10 patients received ZP4207 treatment and 12 patients received Lilly Glucagon treatment in a crossover design. Results are presented by treatment received. Only Part 1 of the trial was conducted.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, ZP4207: In Part 1, 10 patients received treatment with ZP4207 (dasiglucagon) {experimental drug} in the iPhone-based Bionic Pancreas with insulin lispro according to a pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
- Part 1, Lilly Glucagon: In Part 1, 12 patients received treatment with Lilly glucagon in the iPhone-based Bionic Pancreas with insulin lispro according to a pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
Participants
  Participants with AEs | 8 | 12
  Participants with antibodies | 0 | 0
  Participants with edema infusion site reactions | 0 | 0
  Participants with erythema infusion site reactions | 0 | 0
  Participants with investigations AEs | 2 | 2
  Participants with erythrocytes <LLN | 0 | 1
  Participants with hematocrit <LLN | 0 | 1
  Participants with hemoglobin <LLN | 0 | 2
  Participants with lymphocytes <LLN | 0 | 1
  Participants with infusion site pain (VAS) | 0 | 2
  Participants with nausea (VAS) | 4 | 2
  Participants with vascular disorders | 1 | 1

2. Secondary Outcome: Pain Measured on a Visual Analog Scale (VAS)
Description: The VAS scale was used to measure pain at the end of the visit (16 hours) for patients in both treatment groups. The VAS was a psychometric response scale used to measure subjective characteristics of pain. Patients marked a location on a 0 to 10-cm line that corresponded to the amount of pain being experienced, with low scores (cm) indicating no feelings of pain and high scores (cm) indicating high feelings of pain. Actual values are shown. The maximum value in the Lilly glucagon group was recorded at hour 3.
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
cm
  Baseline | 0.00 (0.00) | 0.01 (0.0029)
  Hour 1 | 0.00 (0.00) | 0.00 (0.00)
  Hour 2 | 0.00 (0.00) | 0.00 (0.00)
  Hour 3 | 0.00 (0.00) | 0.06 (0.202)
  Hour 4 | 0.00 (0.00) | 0.00 (0.00)
  Hour 5 | 0.00 (0.00) | 0.00 (0.00)
  Hour 6 | 0.00 (0.00) | 0.00 (0.00)
  Hour 7 | 0.00 (0.00) | 0.02 (0.058)
  Visit end (16 hours) | 0.00 (0.00) | 0.00 (0.00)

3. Secondary Outcome: Nausea Measured on a Visual Analog Scale (VAS)
Description: The VAS scale was used to measure nausea at the end of the visit (16 hours) for patients in both treatment groups. The VAS was a psychometric response scale used to measure subjective characteristics of nausea. Patients marked a location on a 0 to 10-cm line that corresponded to the amount of nausea being experienced, with low scores (cm) indicating no feelings of nausea and high scores (cm) indicating high feelings of nausea. Actual values are shown. The maximum values in both groups were recorded at hour 6, the start of the exercise period.
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
cm
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Hour 1 | 0.12 (0.379) | 0.00 (0.00)
  Hour 2 | 0.00 (0.00) | 0.00 (0.00)
  Hour 3 | 0.11 (0.348) | 0.04 (0.144)
  Hour 4 | 0.00 (0.00) | 0.00 (0.00)
  Hour 5 | 0.02 (0.063) | 0.09 (0.215)
  Hour 6 | 0.29 (0.917) | 0.18 (0.522)
  Hour 7 | 0.00 (0.00) | 0.00 (0.00)
  Visit end (16 hours) | 0.11 (0.348) | 0.00 (0.00)

4. Secondary Outcome: Glycemic Regulation
Description: Measure glycemic regulation, including hypoglycemia exposure (percent of time spent with continuous glucose monitor [CGM] glucose<60mg/dL)
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time points
Groups:
- Part 1, ZP4207: In Part 1, 10 patients received treatment with ZP4207 (dasiglucagon) {experimental drug} in the iPhone-based Bionic Pancreas with insulin lispro according to pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
- Part 1, Lilly Glucagon: In Part 1, 12 patients received treatment with Lilly glucagon in the iPhone-based Bionic Pancreas with insulin lispro according to pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
percentage of time points | 12.78 (17.262) | 17.60 (14.080)
Statistical Analysis 1: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; A paired t-test or the Wilcoxon signed rank test for comparison of means with normally or non normally distributed residuals, respectively, was used. The Shapiro-Wilk test was used to determine the normality of the residuals for each comparison. The residuals were obtained from an analysis of variance (ANOVA) model with treatment group as the fixed effect. If the p-value of the test was <0.001, the non-parametric method was utilized to analyze the endpoint parameter; Test type: Other — A paired t-test was used for the parametric method to compare patients receiving both treatments. A patient was required to have data for both periods to be included in the pre-specified analysis for a given endpoint. Thus, the 2 patients who withdrew from the trial after the Lilly Glucagon treatment before receiving ZP4207 were not included in the analysis; p = 0.2518, t-test, 2 sided; Mean Difference (Final Values) = -6.90, 95% CI 2-sided [-19.63 to 5.84] — The estimated mean difference is based on the difference between the mean values for 10 patients in the ZP4207 group (12.78) and the matching 10 patients in the Lilly glucagon group (19.67)
Statistical Analysis 2: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; Non-parametric method p-value was from a Wilcoxon signed rank text. The normality of the residuals was assessed using the Shapiro-Wilk test, where the residuals were obtained from an ANOVA model with treatment group as the fixed effect. A patient was required to have data for both periods to be included in the pre-specified analysis for a given endpoint; Test type: Other; p = 0.2500, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -8.02, 95% CI 2-sided [-25.85 to 10.68]

5. Secondary Outcome: Average Percent Glucagon Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump.
Description: Secondary endpoint of bionic pancreas function, presented by treatment group. The analysis of bionic pancreas function endpoints was on an intention-to-treat basis.
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of treatment delivered
Groups:
- Part 1, ZP4207: In Part 1, 10 patients received treatment with ZP4207 (dasiglucagon) {experimental drug} with insulin lispro in the iPhone-based Bionic Pancreas according to a pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  ZP4207 (dasiglucagon): A glucagon analog not yet approved by the FDA. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
Percentage of treatment delivered | 96.73 (4.021) | 97.01 (2.851)
Statistical Analysis 1: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.8508, t-test, 2 sided; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-3.55 to 2.99]
Statistical Analysis 2: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; [analysis description as in outcome 4, analysis 2]; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.03, 95% CI 2-sided [-4.12 to 3.13]

6. Secondary Outcome: Average Percent Insulin Dose Amounts Calculated by the Bionic Pancreas Control Algorithm That Are Successfully Delivered by the Pump.
Description: as for outcome 5
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of treatment delivered
Groups:
- Part 1, Lilly Glucagon: In Part 1, 12 patients received treatment with Lilly glucagon with insulin lispro in the iPhone-based Bionic Pancreas according to a pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
Percentage of treatment delivered | 98.36 (1.114) | 97.73 (2.051)
Statistical Analysis 1: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.1847, t-test, 2 sided; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.36 to 1.62]
Statistical Analysis 2: Comparison: Part 1, ZP4207 vs Part 1, Lilly Glucagon; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.0781, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 3.09]

7. Secondary Outcome: Average Percentage of Time During Which the Bionic Pancreas is Functioning Nominally in All Respects Based on Real-time Continuous Glucose Monitoring (CGM) Data
Description: as for outcome 5
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time functioning nominally
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
percentage of time functioning nominally | 95.41 (1.846) | 94.26 (3.966)

8. Secondary Outcome: Average Percentage of Time During Which the Bionic Pancreas is Functioning Nominally With or Without a New CGM Glucose Reading Captured
Description: as for outcome 5
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time functioning nominally
Groups:
- Part 1, Lilly Glucagon: In Part 1, 12 patients received treatment with Lilly glucagon and insulin lispro in the iPhone-based Bionic Pancreas according to a pre-generated randomization scheme.
  Insulin Lispro: Used to lower blood glucose. Commercially available by prescription and is indicated for patients with T1DM, but not for use in a bionic pancreas. Individualized dose based on metabolic needs and frequent monitoring of blood glucose.
  Glucagon: A hormone normally made by the pancreas to raise blood glucose. Used to treat low blood sugar. Commercially available by prescription and is indicated for patients with T1DM in severe hypoglycemia, but not for use in a BP. Subcutaneous administration in one BP arm.
  iPhone-based bionic pancreas: An experimental device.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
percentage of time functioning nominally | 97.86 (1.125) | 96.31 (3.891)

9. Secondary Outcome: CGM Reliability Index, Calculated as Percentage of Possible Values Actually Recorded by CGM
Description: as for outcome 5
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of recorded values
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
percentage of recorded values | 97.55 (1.219) | 97.94 (1.076)

10. Secondary Outcome: CGM Mean Absolute Relative Difference Versus Time-stamped Blood Glucose (BG) Values From Meter Download
Description: as for outcome 5
Time Frame: 16 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
mg/dL | 12.6 (4.13) | 12.7 (5.43)

11. Secondary Outcome: Number of Patients With Technical Faults Associated With the BP Including Cause and Resolution: Calibration Issues
Description: Technical faults in terms of calibration issues were listed by patient.
Time Frame: 16 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
Participants | 9 | 11

12. Secondary Outcome: Number of Patients With Technical Faults Associated With the BP Including Cause and Resolution: Connectivity Issues
Description: Technical faults related to connectivity issues were listed
Time Frame: 16 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 10 | 12
Participants | 3 | 2

13. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Status
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Change
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: T1-Diabetes Distress Scale
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Problem Areas in Diabetes Survey
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Hypoglycemia Fear Survey
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Impact of Daily Diabetes Demands
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Bionic Pancreas User Opinion Survey
Description: This questionnaire was not assessed as per protocol amendment 7.
Time Frame: Up to 3 months
Population: This questionnaire was not assessed as per protocol amendment 7.
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 50 days
Arm/Group | Part 1, ZP4207 | Part 1, Lilly Glucagon
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 8/10 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, ZP4207 (N=10) | Part 1, Lilly Glucagon (N=12)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 2 (5)
Asthenia (General disorders) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 2 (3) | 1 (1)
White blood cell count increased (Investigations) | 2 (2) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 1 (1) — AEs considered as "blood glucose decreased" were distinct from AEs considered as "hypoglycemia"
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (14) | 9 (20)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02971228/SAP_002.pdf
  • Study Protocol (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02971228/Prot_003.pdf